CLINICAL TRIAL: NCT02708654
Title: Automated Hovering for Congestive Heart Failure Management: (EMPOWER) Electronic Monitoring of Patients Offers Way to Enhance Rehabilitation
Brief Title: Automated Hovering for Congestive Heart Failure Patients
Acronym: EMPOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 824816; 1R01HL128465-01 (NIH)
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure
Keywords: Remote monitoring; Incentives
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Participants will be (1) given an electronic pill bottle for their diuretic and a Bluetooth scale; (2) asked to provide the coordinator with name and contact information of a family member or friend to serve as a support partner; (3) will be assigned a 2-digit number to be used as part of the lottery-based engagement incentives in which eligibility to win will be conditional on medication adherence and registering a weight measurement; and, (4) will determine their preferences for Way to Health platform communication methods during the study.(5) Research coordinators to remotely monitor weight gain thresholds and add alert into the participant's electronic health record for verified weight gain
  Interventions: Behavioral: Electronic pill bottle; Behavioral: Bluetooth scale; Behavioral: Support Partner; Behavioral: Engagement incentives
- Control (No Intervention): Participants will receive usual care.

INTERVENTIONS:
Behavioral: Electronic pill bottle — Participant adherence to their diuretic will be monitored on a daily basis and participants will be contacted if they are non-adherence to this medication
  Arms: Intervention
Behavioral: Bluetooth scale — Participant adherence to stepping on their scale will be monitored on a daily basis and participants will be contacted if they are non-adherent to weighing-in. Participant weight gain will also be monitored, and if weight gain exceeds a specific threshold, the managing physician will be notified through the electronic medical record system. Managing providers will also be sent a weekly report of weight measurements.
  Arms: Intervention
Behavioral: Support Partner — Participants will identify a support partner who will be contacted if the participant is non-adherent to their diuretic and/or weighing-in.
  Arms: Intervention
Behavioral: Engagement incentives — Participants will be entered into a daily lottery, for which their participation is contingent on adhering to their diuretic and to weighing-in on the previous day.
  Arms: Intervention

SUMMARY:
Using a 2-arm, randomized controlled trial (RCT) among CHF patients at the University of Pennsylvania Health System (UPHS), to test the effectiveness of applying automated hovering to improve outcomes among CHF patients at high risk of readmission.

DETAILED DESCRIPTION:
Using a 2-arm, randomized, controlled trial (RCT) among congestive heart failure (CHF) patients at the University of Pennsylvania Health System (UPHS), to test the effectiveness of applying automated hovering to improve outcomes among CHF patients at high risk of readmission. This will leverage the electronic medical record (EMR), the Penn Data Store (an electronic repository that can be used to identify study cohorts), and the NIH-funded Way to Health platform, which provides linkages between home-based remote monitoring devices and a server that can provide automated feedback to patients. The primary outcome will be hospital readmission rate during the 12 months of study enrollment. Secondary outcomes will include cost, medication adherence and death. The investigators will enroll CHF patients discharged from UPHS and randomize them to either: usual care with no additional intervention; or 1) the provision of wireless pill bottles and scales with daily lottery incentives to encourage daily adherence 2) asked to provide the name and contact information of a family member or friend to serve as their support partner 3) have their weights monitored for clinically significant threshold, with verified weight gains alerts sent to the managing physician through the EMR. Managing providers will also be sent a weekly report of all weight measurements from the electronic scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a recent University of Pennsylvania Health System hospital (UPHS) discharge of congestive heart failure (CHF) aged 18-80 who will receive follow-up in a UPHS outpatient clinic.

Exclusion Criteria:

* Patients will be excluded if they will not or cannot give consent or have a markedly shortened life expectancy (listed for heart transplant,have a ventricular assist device, are inotrope dependent, metastatic cancer, or dementia)
* end-stage renal disease (since they may not produce urine and be responsive to diuretics).
* on dialysis
* Heart failure managed with a CardioMEMS monitor
* Receiving another remote monitoring/telemedicine intervention
* Receiving follow up care outside of UPHS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2016-05-22 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital readmission rate | 12 months
  Our primary outcome is time to readmission for any cause.The primary comparison will be the times to events compared between the intervention arm and the usual care arm; that is, the primary hypothesis is whether a series of interventions, adapted to the behavior and outcomes of each particular patient, will reduce readmission rates compared to usual care.

SECONDARY OUTCOMES:
Cost | 12 months
  To assess the cost-effectiveness of the intervention, the investigators will use analytic methods for economic evaluations in clinical trials.
Medication adherence to diuretic as measured by electronic pill bottle | 12 months
  Days adherent to medication adherence to diuretic, as measured by electronic pill bottle
Deaths | 12 months
  Deaths

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Only aggregate data will be shared, not on individual level

REFERENCES:
- [Derived] Klaiman T, Iannotte LG, Josephs M, Russell LB, Norton L, Mehta S, Troxel A, Zhu J, Volpp K, Asch DA. Qualitative analysis of a remote monitoring intervention for managing heart failure. BMC Cardiovasc Disord. 2023 Sep 7;23(1):440. doi: 10.1186/s12872-023-03456-9. PMID 37679712
- [Derived] Klaiman T, Ianotte LG, Josephs M, Russell LB, Norton L, Mehta S, Troxel A, Zhu J, Volpp K, Asch D. Qualitative Analysis of a Remote Monitoring Intervention for Managing Heart Failure. Res Sq [Preprint]. 2023 Jan 20:rs.3.rs-2206783. doi: 10.21203/rs.3.rs-2206783/v1. PMID 36712044
- [Derived] Asch DA, Troxel AB, Goldberg LR, Tanna MS, Mehta SJ, Norton LA, Zhu J, Iannotte LG, Klaiman T, Lin Y, Russell LB, Volpp KG. Remote Monitoring and Behavioral Economics in Managing Heart Failure in Patients Discharged From the Hospital: A Randomized Clinical Trial. JAMA Intern Med. 2022 Jun 1;182(6):643-649. doi: 10.1001/jamainternmed.2022.1383. PMID 35532915
- [Derived] Russell LB, Norton LA, Pagnotti D, Sevinc C, Anderson S, Finnerty Bigelow D, Iannotte LG, Josephs M, McGilloway R, Barankay I, Putt ME, Reese PP, Asch DA, Goldberg LR, Mehta SJ, Tanna MS, Troxel AB, Volpp KG. Using Clinical Trial Data to Estimate the Costs of Behavioral Interventions for Potential Adopters: A Guide for Trialists. Med Decis Making. 2021 Jan;41(1):9-20. doi: 10.1177/0272989X20973160. Epub 2020 Nov 20. PMID 33218296
- [Derived] Mehta SJ, Volpp KG, Asch DA, Goldberg LR, Russell LB, Norton LA, Iannotte LG, Troxel AB. Rationale and Design of EMPOWER, a Pragmatic Randomized Trial of Automated Hovering in Patients With Congestive Heart Failure. Circ Cardiovasc Qual Outcomes. 2019 Apr;12(4):e005126. doi: 10.1161/CIRCOUTCOMES.118.005126. PMID 30939922